CLINICAL TRIAL: NCT07189351
Title: Comparative Effects of Muscle Energy Technique and Bowen Therapy on Pain, Range of Motion, and Functional Disability in Patients With Text Neck Syndrome
Brief Title: Comparing Muscle Energy Technique and Bowen Therapy for Pain, Movement, and Disability in Text Neck Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Aqsa Majeed, Dr.Aqsa Majeed, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Asma
Record Dates: First submitted 2025-08-28; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Text Neck Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bowen Therapy with Hot Pack (Experimental): Participants in this group received a hot pack followed by Bowen Therapy in prone lying position. Treatment was administered on alternate days for 6 weeks, with each session lasting 15-20 minutes. Assessments were performed at baseline, week 3, and week 6, with a follow-up at 3 weeks post-treatment.
  Interventions: Other: Bowen Therapy; Other: Muscle Energy Technique (Post-Isometric Relaxation)
- Muscle Energy Technique with Hot Pack (Experimental): Participants in this group received a hot pack applied to the neck and upper back area for 7-10 minutes, followed by Muscle Energy Technique (Post-Isometric Relaxation) for the upper trapezius, levator scapulae, scalenus, and sternocleidomastoid muscles in supine lying position. Each contraction lasted 5 seconds followed by 3 seconds of relaxation, with 5 repetitions per muscle. Treatment was given on alternate days for 6 weeks, with assessments at baseline, week 3, and week 6, and a follow-up after 3 weeks.
  Interventions: Other: Bowen Therapy; Other: Muscle Energy Technique (Post-Isometric Relaxation)

INTERVENTIONS:
Other: Bowen Therapy — Participants received a hot pack, followed by Bowen Therapy performed in prone lying position on a plinth. Bowen moves were applied to soft tissues and muscles of the neck and upper back, aiming to reduce muscle tension and pain. Sessions lasted 15-20 minutes, administered on alternate days for 6 weeks. Assessments were conducted at baseline, 3rd week, 6th week, and at 3-week follow-up.
Other: Muscle Energy Technique (Post-Isometric Relaxation) — Participants received a hot pack applied over the neck and upper back area for 7-10 minutes, followed by Muscle Energy Technique in supine lying position. Post-isometric relaxation was used for upper trapezius, levator scapulae, scalenus, and sternocleidomastoid muscles. A moderate isometric contraction was held for 5 seconds, followed by 3 seconds of relaxation, with 5 repetitions per muscle. Sessions were given on alternate days for 6 weeks. Assessments were performed at baseline, 3rd week, 6th week, and at 3-week follow-up.

SUMMARY:
This study compared the effects of Muscle Energy Technique and Bowen Therapy on patients with Text Neck Syndrome's pain, function ROM, and posture. Today, text neck syndrome is a growing issue. The majority of us experience this unpleasant condition to some extent. There is no study that has compared the effects of muscle energy technique and Bowen therapy, although they can both be quite effective in helping individuals with text neck syndrome reduce their discomfort, improve their range of motion, and improve their functional impairment. So, the goal of this study was to compare the two treatments' results in order to determine whether one was a better method for treating text neck syndrome patients' discomfort by enhancing range of motion and functional impairment.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18-35 years

  * Both genders
  * Using smart phone more than 4 hours per day and pain from last 6 months.
  * Neck disability index greater than 10. (Seemal et al., 2022)

Exclusion Criteria:

* • Subjects who had signs of recent surgery.

  * Whiplash injury or open wounds.
  * Cervical spine pathologies like radiculopathies, disc herniation, spondylolisthesis, sensory changes in neck region..
  * Deformities like torticollis.
  * Any inflammatory or malignant type of pain.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disability | Baseline, 3rd week, 6th week, and 3-week follow-up after treatment completion
  Neck disability Index scale (NDI-U) This Neck Disability Index (NDI) scale assesses the degree of perceived pain in neck an the disability status based on daily activities and underlying cervical spine pain. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. Points summed to a total score